CLINICAL TRIAL: NCT00570804
Title: Oral Cancer Risk Reduction Through Combined Treatment for Tobacco and Alcohol Use
Brief Title: Combined Treatment for Tobacco and Alcohol Use in Puerto Rico
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2005-0791; U54CA096300 (NIH); U54CA096297 (NIH); NCI-2012-02110 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2007-12-07; First posted 2007-12-11 (Estimated); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Smoking
Keywords: Smoking Cessation; Puerto Rico Quitline; Motivational Relapse Prevention; Oral Cancer; Risk Reduction; Tobacco Use; Alcohol Use; MAPS; Motivation and Problem-Solving; Telephone Interview; Counseling
MeSH Terms: conditions — Smoking; Smoking Cessation; Mouth Neoplasms; Risk Reduction Behavior; Tobacco Use; Alcohol Drinking | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MAPS+ (Other): MAPS+ (Motivation and Problem-Solving Plus):
  Counseling using specific treatment approach that focuses on combined smoking cessation and the reduction of at-risk alcohol use.
  Interventions: Behavioral: Telephone Counseling; Behavioral: Telephone Assessments
- MAPS (Other): MAPS (Motivation and Problem-Solving):
  Counseling treatment approach with a focus on smoking cessation.
  Interventions: Behavioral: Telephone Counseling; Behavioral: Telephone Assessments

INTERVENTIONS:
Behavioral: Telephone Counseling — 7 counseling calls where quit date set on first counseling call; then counseling calls on quit date, 3-5 days after quit date, 7-10 days after quit date, 15-30 days after quit date, 45-60 days after quit date, and 90 days after quit date, each taking about 15 to 30 minutes to complete.
Behavioral: Telephone Assessments — 4 assessment telephone calls at Weeks 12, 26 and 52 (interview by a research staff member), taking about 30 minutes each to complete.
  Other Names: Survey; Questionnaire

SUMMARY:
Objectives:

1. Assess MAPS and MAPS+ effects on alcohol at-risk behaviors and smoking cessation.
2. Assess MAPS and MAPS+ effects on treatment mechanisms (increased self-efficacy, decreased temptations/craving, decreased stress and negative affect) and the role of those mechanisms in mediating MAPS and MAPS+ effects on alcohol at-risk behaviors and smoking cessation.
3. Evaluate the cost-effectiveness of MAPS and MAPS+ in the reduction of at-risk drinking and smoking cessation.

DETAILED DESCRIPTION:
Participants for this study will be recruited mainly through media advertisements (such as TV, radio, newspapers, magazines, etc.).

If you are interested in participating in this study, you will be asked to provide demographic information, such as your name, telephone number, and address. You will then be mailed a packet, which will include a copy of this informed consent document, self-help reading materials, and a guide to answering the questionnaires.

Within about 2 weeks after you have received your packet, you will be interviewed by a research staff member by phone. You will be given detailed information about this study as part of the consent process. This is a telephone counseling study. Please read this copy of the consent very carefully. When the research staff member calls you in about 2 weeks, he or she will review this consent form with you. You should ask any questions you have about the consent or the study, and discuss any concerns you have with the research staff member. After discussing the consent and the study with the research staff member, you will be asked if you have read and understood the consent, and asked if you agree to participate in this study. Your consent to participate in this study will be tape recorded. This is so researchers can verify (know) that you have freely consented to participating in this study. You should keep this copy of the consent, and you may ask questions about it and/or the study at any time.

If you agree to participate, you will then go over several questionnaires with the interviewer. You may be asked questions about your living situation, mood, depression, anxiety, sleeping habits, appetite, smoking and alcohol use habits, social status, finances, job, physical activity, and support base (family and/or friends). Then a quit date will be set as well as the first telephone counseling call. This interview may take a total of about 1 hour to complete.

After this interview, participants will be randomly picked (as in the toss of a coin) to be in one of 2 groups. One group will receive standard quit-smoking counseling to help decrease their risk of cancer. The other group will also receive counseling, which will focus on decreasing the risk of getting cancer by decreasing smoking and alcohol use.

Your counselor will be contacting you to set up your first counseling call. You will receive a total of 7 counseling calls. You will discuss the timing of the counseling calls with your counselor based upon when it is felt to be most beneficial for you. Depending on which group you are in, you will be counseled on strategies for quitting smoking and/or decreasing alcohol use to help decrease your risk of cancer. These calls will take about 15 to 30 minutes each to complete.

At Weeks 12, 26 and 52, you will be interviewed by telephone by a research staff member, who will cover the same information as before. These evaluation (assessment) calls will take about 30 minutes each to complete. You will receive a total of 4 assessment phone calls. You will receive a total of 11 calls (including the counseling and assessment calls) over about a 12-month period of time.

Your counseling calls (not the assessment calls) will be tape recorded. You will be reminded before each counseling call that it will be taped recorded. This is so researchers can make sure that correct procedures are being followed. Only the study staff will be allowed to listen to these tapes. Your identity will be kept secure and confidential. These tapes will be erased when this study has ended.

Your participation in this study will be over after the assessment call at Week 52.

This is an investigational study. Up to 370 participant will take part in this multicenter study. None will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Current (daily) smoker requesting help for smoking cessation
2. Exhibit at least one of the following criteria for at-risk drinking: a) an average of =/> 2 alcoholic beverages/day during the past 30 days for men or =/>1 drink/day for women, OR b) two or more occasions of consuming /=> 5 alcoholic beverages during the past 30 days for men or =/>4 drinks for women, OR c) in the past 30 days, driving after consuming =/>3 drinks.
3. Age 18 or above
4. Motivated to quit smoking in the next 30 days
5. Viable (working) telephone number and home address
6. No other household member enrolled in this protocol
7. Residing in Puerto Rico
8. Must score less than or equal to 15 on the AUDIT (Alcohol Use Disorders Identification Test)

Exclusion Criteria:

1. Currently incarcerated or in jail
2. Currently pregnant
3. Score equal to or more than 16 on the Alcohol Use Disorders Identification Test (AUDIT) measure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 370 (Estimated)
Dates: Start 2007-12 (Actual); Primary Completion 2021-07-22 (Actual); Study Completion 2021-07-22 (Actual)

PRIMARY OUTCOMES:
Continuous outcome variables (including number of drinks per day, self-efficacy, etc.) | 2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Lorna McNeill, MPH,PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org